CLINICAL TRIAL: NCT03830268
Title: Optimisation of Acute Medium Chain Triglycerides Intake Characteristics on Different Plasma Metabolites in Young and Older Participants
Brief Title: Acute Medium Chain Triglycerides (MCT) Intake in Young and Older Participants
Acronym: Opti-MCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2017-714
Record Dates: First submitted 2019-02-01; First posted 2019-02-05 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Ketonemia
Keywords: Ketones; Medium Chain Triglycerides; Glucose; Insulin; Free fatty acids
MeSH Terms: conditions — Ketosis; Insulin Resistance | interventions — Breakfast; Lunch

STUDY DESIGN:
Intervention Model Description: 10 young and 10 older participants undergoing six separate but identical metabolic visits (interventions)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MCT intake in young participants (Experimental): Different conditions paired with a dietary MCT beverage over an 8-hour metabolic day protocol in young participants.
  Interventions:
  1. No MCT intake with breakfast, no lunch (i.e. CTL)
  2. No MCT intake with lunch, no breakfast (i.e CTL inverted)
  3. 10g of Betaquik with breakfast, no lunch (i.e BQ10)
  4. 20g of Betaquik with breakfast, no lunch (i.e BQ20)
  5. 10g of Betaquik with low-carbs breakfast, no lunch (i.e BQ10LC)
  6. 10g of Betaquik with lunch, no breakfast (i.e BQ10 inverted)
  Interventions: Dietary Supplement: No MCT intake with breakfast, no lunch; Dietary Supplement: No MCT intake with lunch, no breakfast; Dietary Supplement: 10g of Betaquik; Dietary Supplement: 10g of Betaquik with low-carbs breakfast; Dietary Supplement: 20g of Betaquik; Dietary Supplement: 10g of Betaquik with lunch, no breakfast
- MCT intake in older participants (Experimental): Different conditions paired with a dietary MCT beverage over an 8-hour metabolic day protocol in older participants.
  Interventions:
  1. No MCT intake with breakfast, no lunch (i.e. CTL)
  2. No MCT intake with lunch, no breakfast (i.e CTL inverted)
  3. 10g of Betaquik with breakfast, no lunch (i.e BQ10)
  4. 20g of Betaquik with breakfast, no lunch (i.e BQ20)
  5. 10g of Betaquik with low-carbs breakfast, no lunch (i.e BQ10LC)
  6. 10g of Betaquik with lunch, no breakfast (i.e BQ10 inverted)
  Interventions: Dietary Supplement: 10g of Betaquik

INTERVENTIONS:
Dietary Supplement: No MCT intake with breakfast, no lunch — Water given with a regular standardize breakfast and water given at noon without lunch.
  Other Names: CTL
  Arms: MCT intake in young participants
Dietary Supplement: No MCT intake with lunch, no breakfast — Water given in the beginning of the metabolic study day without breakfast and water given at noon with a regular standardize lunch.
  Other Names: CTL inverted
  Arms: MCT intake in young participants
Dietary Supplement: 10g of Betaquik — BQ10 given with a regular standardize breakfast and BQ10 given at noon without lunch.
  Other Names: BQ10
Dietary Supplement: 10g of Betaquik with low-carbs breakfast — BQ10 given with a low-carbs standardize breakfast and BQ10 given at noon without lunch.
  Other Names: BQ10LC
  Arms: MCT intake in young participants
Dietary Supplement: 20g of Betaquik — BQ20 given with a regular standardize breakfast and BQ20 given at noon without lunch.
  Other Names: BQ20
  Arms: MCT intake in young participants
Dietary Supplement: 10g of Betaquik with lunch, no breakfast — BQ10 given in the beginning of the metabolic study day without breakfast and BQ10 given at noon with a regular standardize lunch.
  Other Names: BQ10 inverted
  Arms: MCT intake in young participants

SUMMARY:
Compare plasma metabolites following different conditions paired with a dietary MCT beverage over an 8-hour metabolic day protocol in young and older participants.

ELIGIBILITY:
Inclusion Criteria:

* 10 health young (20-40 y old) and 10 health older (> 60 y old) participants
* Men and women

Exclusion Criteria:

* smoking
* diabetes (fasting glucose >7.0 mmol/l and glycated hemoglobin >6.9%)
* strenuous aerobic exercise more than three times a week
* untreated hypertension, dyslipidemia, and abnormal renal, liver, heart or thyroid function
* under medication known to affect triglycerides and carbohydrates metabolism (i.e. diuretics, beta-blockers, steroids, insulin sensitizing)

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-06-02 (Actual); Primary Completion 2019-06-25 (Actual); Study Completion 2019-06-25 (Actual)

PRIMARY OUTCOMES:
Concentration of plasma ketones (acetoacetate and B-hydroxybutyrate) | 8 hours
  To compare acute ketonemia following different conditions paired with a dietary MCT beverage over an 8-hour metabolic day protocol.

SECONDARY OUTCOMES:
Concentration of plasma glucose | 8 hours
  To compare acute glucose following different conditions paired with a dietary MCT beverage over an 8-hour metabolic day protocol.
Concentration of plasma insulin | 8 hours
  To compare acute insulin following different conditions paired with a dietary MCT beverage over an 8-hour metabolic day protocol.
Concentration of plasma free fatty acids | 8 hours
  To compare acute free fatty acids following different conditions paired with a dietary MCT beverage over an 8-hour metabolic day protocol.

CONTACTS AND LOCATIONS:
Locations (1):
- Rearsh Centre on Aging, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cunnane SC, Courchesne-Loyer A, St-Pierre V, Vandenberghe C, Pierotti T, Fortier M, Croteau E, Castellano CA. Can ketones compensate for deteriorating brain glucose uptake during aging? Implications for the risk and treatment of Alzheimer's disease. Ann N Y Acad Sci. 2016 Mar;1367(1):12-20. doi: 10.1111/nyas.12999. Epub 2016 Jan 14. PMID 26766547
- [Background] Croteau E, Castellano CA, Fortier M, Bocti C, Fulop T, Paquet N, Cunnane SC. A cross-sectional comparison of brain glucose and ketone metabolism in cognitively healthy older adults, mild cognitive impairment and early Alzheimer's disease. Exp Gerontol. 2018 Jul 1;107:18-26. doi: 10.1016/j.exger.2017.07.004. Epub 2017 Jul 12. PMID 28709938
- [Background] Courchesne-Loyer A, Croteau E, Castellano CA, St-Pierre V, Hennebelle M, Cunnane SC. Inverse relationship between brain glucose and ketone metabolism in adults during short-term moderate dietary ketosis: A dual tracer quantitative positron emission tomography study. J Cereb Blood Flow Metab. 2017 Jul;37(7):2485-2493. doi: 10.1177/0271678X16669366. Epub 2016 Jan 1. PMID 27629100
- [Background] Courchesne-Loyer A, Fortier M, Tremblay-Mercier J, Chouinard-Watkins R, Roy M, Nugent S, Castellano CA, Cunnane SC. Stimulation of mild, sustained ketonemia by medium-chain triacylglycerols in healthy humans: estimated potential contribution to brain energy metabolism. Nutrition. 2013 Apr;29(4):635-40. doi: 10.1016/j.nut.2012.09.009. Epub 2012 Dec 28. PMID 23274095
- [Background] Castellano CA, Nugent S, Paquet N, Tremblay S, Bocti C, Lacombe G, Imbeault H, Turcotte E, Fulop T, Cunnane SC. Lower brain 18F-fluorodeoxyglucose uptake but normal 11C-acetoacetate metabolism in mild Alzheimer's disease dementia. J Alzheimers Dis. 2015;43(4):1343-53. doi: 10.3233/JAD-141074. PMID 25147107